CLINICAL TRIAL: NCT06771817
Title: Feasibility and Preliminary Effectiveness of Written Exposure Therapy (WET) for Pregnant or Postpartum Adolescents and Youth With Post-Traumatic Stress Disorder (PTSD) in an Open Pilot Trial
Brief Title: Empowering Perinatal Adolescents Through Writing
Acronym: EMPWR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Texas Child Mental Healthcare Consortium (TCMHCC) (Unknown)
Responsible Party: Principal Investigator, Nabila Haque, Resident-Psychiatry, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU-2024-1115; NECMHR01-FY24 -060 (Other Grant/Funding Number: Texas Child Mental Healthcare Consortium (TCMHCC))
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Post-Traumatic Stress Disorder in Adolescence; PTSD - Post Traumatic Stress Disorder; PTSD and Trauma-related Symptoms; Pregnancy and PTSD
Keywords: PTSD; post-traumatic stress disorder; post-partum; pregnant; adolescent; adolescent PTSD; trauma; written exposure therapy; therapy; adolescent pregnancy; written exposure
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Written Exposure Therapy (Experimental): All participants will receive written exposure therapy
  Interventions: Behavioral: Written Exposure Therapy

INTERVENTIONS:
Behavioral: Written Exposure Therapy — WET may be an optimal treatment for pregnant or postpartum adolescents and youth with PTSD in a low resource setting. WET addresses many of the barriers above. It is delivered in just 5 sessions, with no homework, and may promote a sense of self-efficacy in adolescents and youth due to the nature of writing assignments and brief therapist involvement. It is attractive in resource-poor settings because just 10-15 min of direct therapist time per follow-up session is needed.

SUMMARY:
This is a feasibility and acceptability study of Written Exposure Therapy (WET) for PTSD in pregnant and postpartum adolescents and youth with PTSD.

DETAILED DESCRIPTION:
The main goal of this research study is to investigate whether a short trauma-focused therapy involving writing is something teens and young adults who are pregnant or recently had a baby and have symptoms related to post-traumatic stress disorder (PTSD) are able to complete. This study is specifically examining the feasibility and acceptability of Written Exposure Therapy (WET) as a treatment in this population. WET is a type of therapy where people write about a traumatic experience they have gone through, and their feelings about the event. Doing this over several sessions may help some people reduce how distressing the memory is to them over time.

In addition, this study aims to investigate if WET can reduce symptoms related to PTSD in teens and young adults who are pregnant or have had a baby in the last year. The study will also explore if it is possible to gather enough information on measurements like heart rate and sleep patterns with smart watches in the same population, to look at brain patterns before and after the therapy, and to see if WET can improve emotions, functioning, and relationships in pregnant and post-partum individuals.

Prior to initiating the course of WET, participants will undergo screening procedures to evaluate eligibility. Those eligible will complete 5 sessions of written exposure therapy, one session per week and biomarker data will be collected via a wearable device. Participants will also undergo optional electroencephalography (EEG) as well as self-report and clinician-rated assessments. Follow-up visits will be conducted at 4, 8 and 12 weeks post-baseline (post-treatment for WET), with weekly assessments.

The baseline visit must be done in-person in order to set up the smart watch. If participants choose to undergo electroencephalography, they will be required to come in-person for the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Have been referred by a clinician to the study or receiving standard of care treatment for pregnancy or post-partum follow-up
3. Aged 15-24 at time of screening
4. Either have Gestational age >12 weeks or be <1 year postpartum at time of screening
5. Able and willing to provide informed consent if 18 years of age or above or the legal guardian must be able and willing to provide informed consent if participant is less than 18 years of age and participant willing and able to provide assent if less than 18 years of age
6. Able to read, write and speak in English and Spanish; if the participant is under age 18, parents must be able to understand spoken or written English or Spanish.
7. Have the ability to complete clinical evaluations and self-report measures.
8. Meet diagnostic or subthreshold criteria for PTSD.

Exclusion Criteria:

1. Have any condition for which, in the opinion of the investigator or designee, study participation would not be in their best interest (including but not limited to cognitive impairment, unstable general medical condition, intoxication, active psychosis) or that could prevent, limit, or confound the protocol-specified assessments.
2. Have current mania, hypomania, or psychosis
3. Be at serious suicidal risk that cannot be managed in the outpatient setting
4. Pervasive or intellectual developmental disorder requiring substantial or very substantial support.
5. Currently receiving or having received course of exposure-based therapy (e.g. WET, PE, CPT, or TF-CBT) in the past six months

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Written Exposure Therapy | From enrollment to study exit visit at week 12
  Feasibility will be assessed based on recruitment, retention and treatment adherence rates. Acceptability will be evaluated through participant feedback, including satisfaction with the intervention and willingness to engage in treatment. The primary outcome will be the percentage of participants who complete treatment within 4 weeks, for a 12-week study period. We expect at least 70% of participants will be able to complete treatment within 4 weeks.

SECONDARY OUTCOMES:
Changes in PTSD Symptom Severity Assessed by the Clinician Administered Scale for PTSD (CAPS-5) | From enrollment to study exit visit at week 12
  The Clinician-Administered PTSD Scale for DSM-5 - Child/Adolescent Version (CAPS-CA-5) is a 30-item clinician-administered PTSD scale based upon DSM-5 criteria for children and adolescents ages 7 and above. It is a modified version of the CAPS-5 that includes age-appropriate items and picture response options. It will be used to diagnose PTSD or subthreshold PTSD and obtain data on the frequency and severity of PTSD symptoms. The worst traumatic event identified in the LSC-R from baseline will be used for all CAPS-CA-5 administrations. Preliminary effectiveness will be measured by assessing changes in the CAPS-5 score at 4,8, and 12 weeks after baseline visit.
Changes in PTSD Symptoms Assessed by the PTSD Checklist for DSM-5 | From enrollment to study exit visit at week 12
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Scores range from 0 to 80 and a score above 21 is indicative of probable PTSD. A 10-20 point change represents clinically significant change.
Change in Sleep Quality Assessed by the Pittsburgh Sleep Quality Index (PSQI) | From enrollment to study exit visit at week 12
  Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report measure to evaluate sleep quality, duration, and functioning.
Changes in Emotional Regulation Assessed by the Difficulties in Emotion Regulation Scale (DERS-16) | From enrollment to study exit visit at week 12
  The Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) is a 16-item assessment of emotion regulation difficulties, rated on a 5-point Likert scale.
Changes in Anxiety Assessed by the Perinatal Anxiety Screening Scale (PASS) | From enrollment to study exit visit at week 12
  The Perinatal Anxiety Screening Scale (PASS) is a 31-item self-rated questionnaire investigating anxiety symptoms during the last month in child-bearing women. Scores may range 0-93 and cutoff for clinical anxiety is ≥26.

CONTACTS AND LOCATIONS:
Overall Officials: Nabila Haque, MD., PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Center for Depression Research and Clinical Care, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmadi SJ, Musavi Z, Samim N, Sadeqi M, Jobson L. Investigating the Feasibility, Acceptability and Efficacy of Using Modified-Written Exposure Therapy in the Aftermath of a Terrorist Attack on Symptoms of Posttraumatic Stress Disorder Among Afghan Adolescent Girls. Front Psychiatry. 2022 Apr 8;13:826633. doi: 10.3389/fpsyt.2022.826633. eCollection 2022. PMID 35463492
- [Background] Nillni YI, Baul TD, Paul E, Godfrey LB, Sloan DM, Valentine SE. Written exposure therapy for treatment of perinatal PTSD among women with comorbid PTSD and SUD: A pilot study examining feasibility, acceptability, and preliminary effectiveness. Gen Hosp Psychiatry. 2023 Jul-Aug;83:66-74. doi: 10.1016/j.genhosppsych.2023.04.013. Epub 2023 Apr 24. PMID 37119780